CLINICAL TRIAL: NCT04163796
Title: Evaluation of an Upright Powered Wheelchair for People With SCI
Brief Title: UPnRIDE Power Standing Wheelchair for SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx Veterans Medical Research Foundation, Inc (Other)
Responsible Party: Principal Investigator, EunKyoung Hong, Postdoctoral Researcher, Bronx Veterans Medical Research Foundation, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SPU-17-036
Record Dates: First submitted 2018-06-18; First posted 2019-11-15 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- UPnRIDE Training (Experimental): During each session, heart rate (HR), blood pressure (BP), total session time, time in standing posture, count of sit-to-stand positioning, total distance of overground movement, and rating of perceived exertion (Borg scale) for mobility skills will be monitored. At all study visits during the training period, participants will be asked to answer general health questions about the occurrence of any pressure ulcers or infections.
  Interventions: Device: UPnRIDE power wheelchair

INTERVENTIONS:
Device: UPnRIDE power wheelchair — The intervention will consist of approximately 3.5 hours per session, 3 times per week over 12 weeks. During each 3.5-hour session, subjects will be asked to stand at least 5 minutes during every 15 minutes or more as tolerated. One time each session, participants will be asked to perform the Activities of Daily Living course.

SUMMARY:
People with higher level of spinal cord injury have limitations to using exoskeletal-assisted walking devices due to restrictions of trunk stability, functional use of the upper extremities and hand grip. With increasing sedentary time in wheelchairs, people with SCI have a high risk for developing secondary complications. A powered wheelchair has recently been developed for use in persons with spinal cord injury that provides a solution for placing the user in an upright, standing position while maintaining the overground mobility features of the powered wheelchair; providing the ability to engage in society in either a standing or seated position. The purpose of this study is to verify user performances of the upright powered wheelchair and to identify obstacles that are difficult, or prevent use. Additionally, the option to have upright posture throughout the day may have the potential to improve some of the secondary medical conditions associated with the extreme sedentary lifestyle.

This study will determine change from baseline after 12 weeks of use for safety, tolerance, medical, physical and quality of life outcomes. The intervention will consist of 3.5 hours per session, 3 times per week for 12 weeks. During each session, participants will be asked to stand at least 5 minutes during every 15 minutes. To our knowledge, there is no existing empirical data on intermittent standing during the day in persons with higher levels of SCI who cannot otherwise stand and whether this approach will improve health related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Power wheelchair user as a primary means of mobility;
2. 18-89 years old;
3. ≥1 year after SCI;
4. Height of 160 to 190 cm;
5. Weight of <100 kg; and
6. Able to sign informed consent.

Exclusion Criteria:

1. Able to ambulate with or without an assistive device or physical assistance greater than 4 consecutive steps;
2. Any pressure ulcer at any body location that is deemed to be contraindicated for a power wheelchair or standing frame by the study physician;
3. Concurrent medical disease that would be exclusionary for standing (as per the clinical judgment of the study physician);
4. Severe spasticity (Ashworth 4) or uncontrolled clonus;
5. History of fragility fractures, long bone fractures in the past 1 years, heterotrophic ossification, or other bone conditions that would be exclusionary for use of a standing modality as per the clinical judgment of the study physician;
6. Significant contractures that would be exclusionary for use of a standing modality as per the clinical judgment of the study physician
7. Psychiatric or cognitive status that may interfere with the ability to follow instruction to use the device; and
8. Pregnant or lactating women.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Wheelchair mobility skills - RPE | Training Period - 36 Sessions up to 12 weeks
  Participants will be requested to perform a rating of perceived exertion (RPE).
Wheelchair mobility skills - FIM | Training Period - 36 Sessions up to 12 weeks
  Participants will be requested to perform a rating Functional Independence Measurement (FIM) for each UPnRIDE activity.
Activities Daily Living Course - RPE | Training Period - 36 Sessions up to 12 weeks
  Participants will be requested to perform a rating of perceived exertion (RPE) during the Activities Daily Living Course (ADLC).
Activities Daily Living Course - FIM | Training Period - 36 Sessions up to 12 weeks
  Participants will be requested to perform a rating Functional Independence Measurement (FIM) during the Activities Daily Living Course (ADLC).

SECONDARY OUTCOMES:
Postural orthostatic hypotension blood pressure tolerance test (OH BP) | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  Participants will be in the supine position on a bed or elevated gym mat and beat-to-beat HR will be recorded for 60 seconds, followed by passive re-positioning to the seated position on a bed or elevated gym mat with the hip and knee at a 90° angle and the lower leg hanging off the side. Passive repositioning will be accomplished by one staff member lifting the participant's torso by the shoulders, while supporting the head and neck, and a second staff member shifting the subject perpendicular to the bed and allowing the participant's legs to hang off the side. Participants will be instructed not to assist in the passive movement during this transition, and will be supported by staff.
Pulmonary function tests - Spirometry | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  While seated in the chair and after a mouth piece and nose clip are applied, the subject will be asked to breathe normally for 3 to 6 breaths. They will then be instructed to forcibly inhale until their lungs are filled. After a brief pause, they will then be instructed to forcibly exhale the air in their lungs and hold the maneuver for approximately 6 seconds. After a brief rest, the maneuver will be repeated a minimum of three times to ensure reliability.
Pulmonary function tests - Static Lung Volumes | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  The volume of air in the lungs will be assessed using the nitrogen washout technique. The nitrogen washout technique, which takes about five minutes to perform, will begin while a subject is seated in his/her wheelchair and after a mouth piece and nose-clips have been applied. The subject will then be asked to breathe room air into and out of the mouthpiece for 3-6 breaths. The air exhaled, which normally contains mostly nitrogen, will be collected and analyzed by the pulmonary function cart. Once a participant has completed the 3-6 breaths, s/he will be asked to take a slow deep breath in and to exhale until the lungs are empty, after which the participant returns to a normal breathing pattern. Following an additional 3-6 regular breaths, the pulmonary function cart will begin delivering 100% oxygen through the mouthpiece. The subject will continue to inhale 100% oxygen while taking normal breaths until oxygen is the only gas measurable in his/her exhaled air.
Pulmonary function tests - Breathing Pattern | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  Resting breathing pattern will be measured by abdominal and thoracic respiratory inductive plethysmography. The participant will be asked to wear two chest straps for a designated period of time. Signals from the participant's chest wall excursions are analyzed for indices of resting breathing pattern such as tidal volume and timing and derivatives of these measurements.
Inflammatory biomarkers | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  Due to its clinical utility and widespread use to measure risks for coronary heart disease, the primary outcome assessment of systemic inflammation will be levels of CRP, which will be measured in sera using a commercially available ELISA. Additional exploratory analyses may be performed using commercially available single- and multi-plex immunoassays to assay the following: HMGb1, IL-1β, IL-1Ra, IL-6, IL-8, IL-10, IL-15, MIF, MIP1-α/CCL3, TNF-α, leptin, and adipokine.
Body Composition | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  A dual energy x-ray absorptiometry (DXA) scan for regional and total body fat, lean and bone tissue masses will be performed two times: at baseline and post.
Bowel function surveys - 10Q Bowel Function Survey (BFS) | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  The 10Q Bowel Function Survey (BFS) will be administered three times: at baseline, midpoint, and post.
Bowel function surveys - Bristol Stool Scale | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  The Bristol Stool Scale (BSS) will be administered three times: at baseline, midpoint, and post. The BSS is a diagnostic medical tool designed to classify the form of human faces into seven categories (Type 1 to 7: Hard lumps to Soft/Liquid).
SCI-QOL | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  The Spinal Cord Injury Quality of Life measurement tool is the first validated SCI-specific QOL measurement tool for the field. The specific short form item banks to be use are: Bowel and Bladder Management Difficulties from the Physical Medical Domain, Ability to Participate and Independence from the Social Domain, and Positive Affect, and Resilience from Emotional Domain. These will be performed three times: at baseline, midpoint, and post.
Lipid Profile - Cholesterols | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  Total cholesterol (TC), low density lipoprotein cholesterol (LDL-c), triglyceride (TG) and high density lipoprotein cholesterol (HDL-c) values will be measure and samples will be collected at baseline, midpoint and post.
Homeostatic Model of Insulin Resistance (HOMA-IR) | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  The standard equation for the HOMA-IR will be used to calculate insulin resistance [HOMA-IR = FPG (mg/dl) x FPI(μU/mL) / 405].
Serum total testosterone levels | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  Serum total testosterone will be determined by a radioimmunoassay (RIA; MP Biomedicals, Costa Mesa, CA) kit with an intra-assay CV of 10.0, 9.6, and 13% at 1.4, 4.6, and 8.0 nmol/L41,61,62. Measurements will be performed pre, midpoint and post.
Serum estradiol levels | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  Serum estradiol values will be determined by a commercial kit assay using RIA (MP Biomedicals, Costa Mesa, CA) with an intra-assay CV of 15.7, 5.5, and 3.5% at 25.4, 152, and 657 pg/mL63. Measurements will be performed pre, midpoint and post.
Lower extremity blood flow | Evaluations - Baseline/After session 18 (up to 6 weeks) /After session 36 (up to 12 weeks)
  Lower extremity blood flow will be measured by strain gauge and will be assessed at sessions 1 and 36.

CONTACTS AND LOCATIONS:
Overall Officials: EunKyoung Hong, PhD, Principal Investigator — Bronx VMRF
Locations (1):
- Spinal Cord Damage Research Center, The Bronx, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT04163796/ICF_000.pdf